CLINICAL TRIAL: NCT06082297
Title: Can Blood Flow Enhancing Plantar Flexion Electrically Induced Via Textile Electrodes in a Sock Using 1 Hz Frequency Give Better Comfort and Energy Efficiency as Compared to 36 Hz ?
Brief Title: Evaluation in 15 Participants of Blood Flow, Comfort and Efficiency, Using 1 vs 36 Hz Stimulation Via Textile Electrodes
Acronym: TTE_PVV_1_36
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Professor,MD,PhD, Karolinska University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TTE_PVV_1_vs_36_Hz
Record Dates: First submitted 2023-09-30; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Hemodynamic Instability; Pain
Keywords: Neuromuscular electrical stimulation; Hemodynamics; Physical inactivity
MeSH Terms: conditions — Pain; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Repeated measures tests on on each of the 15 participants, comparing outcomes for no intervention and 10 different interventions in the form of variations in parameter-settings of neuromuscular electrical stimulation, with gradually increasing current amplitude until induction of ankle plantar flexion.
Masking Description: Participants did not receive information about what parameter-settings that were used for the different tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where repeated measures where performed in 15 participants. (Experimental): Each of the 15 participants in the arm was, in addition to the resting state (no intervention), exposed to 10 different interventions repeated after each other to enable repeated measures of the outcomes.
  Interventions: Device: Chattanooga Physio, DJO, neuromuscular electrical stimulation

INTERVENTIONS:
Device: Chattanooga Physio, DJO, neuromuscular electrical stimulation — Neuromuscular electrical stimulation (NMES) was applied with a device called Chattanooga Physio (DJO), testing 10 different combinations of parameter-settings. The parameter-settings that were varied and combined were frequency (1Hz and 36Hz) and plateau times (0.5s, 1.5s, 3s, 5s, 7s). The NMES was applied to the calf of the participants via transversally placed textile electrodes (3x3 cm) integrated in a sock starting with very low current amplitude followed by gradual small increases in current amplitude until induction of ankle plantar flexion, at which time-point the outcomes where measured.
  Other Names: Device name and manufacturer:

SUMMARY:
Muscle contractions induced by calf low-intensity neuromuscular electrical stimulation (C-LI-NMES) can increase venous return and may reduce venous thromboembolism. This study aimed to compare the effect of different C-LI-NMES frequencies and plateau times on hemodynamics, discomfort and energy efficiency, when applied via sock-integrated transverse textile electrodes.

DETAILED DESCRIPTION:
Fifteen healthy participants were stimulated via two 3x3cm transverse textile electrodes integrated in a sock, with ten different combinations of frequency (1Hz or 36Hz) and plateau times (0.5/1.5/3/5/7s), with gradually increasing NMES-intensity until plantar flexion-induction. At this point, popliteal peak venous velocity (PVV), time-averaged mean velocity (TAMV) and ejection volume (EV) were assessed by Doppler-ultrasound, discomfort by a numerical rating scale (NRS, 0-10) and values for current amplitude and energy were calculated based on the NMES-device´s intensity level. Values expressed with median (interquartile range), significance set to p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99 years of age
* Voluntary participation

Exclusion Criteria:

* Pregnancy
* Pacemaker
* Ongoing thromboprophylaxis
* Skin wounds
* Vascular abnormalities
* Previous vascular system surgery in the lower limbs

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Peak venous velocity (PVV) | Day 1 at rest (baseline, no intervention) and when ankle plantar flexion was induced by the intervention
  Peak venous velocity (centimeters per second) will be assesed by Doppler ultrasound of in the popliteal vein
Time averaged mean velocity (TAMV) | Day 1 at rest (baseline, no intervention) and when ankle plantar flexion was induced by the intervention
  Time averaged mean velocity will be assesed by Doppler ultrasound in the popliteal vein (centimeters per second)
Average duration of blood pulse (ADBP) | Day 1 at rest (baseline, no intervention) and when ankle plantar flexion was induced by the intervention
  Average duration of blood pulse will be assesed by Doppler ultrasound in the popliteal vein (seconds)
Ejection volume (EV) | Day 1 at rest (baseline, no intervention) and when ankle plantar flexion was induced by the intervention
  Ejection volume of blood will be assesed by Doppler ultrasound in the popliteal vein (milliliters)

SECONDARY OUTCOMES:
Numerical rating scale (NRS) | Day 1 during ankle plantar flexion was induced by the intervention
  Discomfort estimated using a numerical rating scale from 0 (no pain) to 10 (worst pain)
Current amplitude | Day 1 during ankle plantar flexion was induced by the intervention
  Current amplitude in milliampere (mA) will be assessed by using stepwise increases (typically 1mA) on the NMES device until a plantar flexion is induced
Energy | Day 1 during ankle plantar flexion was induced by the intervention
  Energy per stimulation cycle in millijoule (mJ) will be assessed by using stepwise increases (typically 1mA) on the NMES device until a plantar flexion is induced, at which point the energy consumption (mJ) is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ackermann, PhD, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska university Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share individual participant data, but individual participant data may be shared upon reasonable request in the future.

REFERENCES:
- [Derived] Juthberg R, Flodin J, Aliaga N, Guo L, Rodriguez S, Persson NK, Ackermann PW. Electrically induced hemodynamic enhancement via sock-integrated electrodes is more comfortable and efficient at 1 hz as compared to 36 hz. Sci Rep. 2025 Apr 15;15(1):12944. doi: 10.1038/s41598-025-97431-3. PMID 40234723